CLINICAL TRIAL: NCT02834403
Title: Clinical Phase Ib/II Trial of L-NMMA Plus Taxane Chemotherapy in the Treatment of Refractory Locally Advanced or Metastatic Triple Negative Breast Cancer Patients
Brief Title: L-NMMA Plus Taxane Chemotherapy in Refractory Locally Advanced or Metastatic Triple Negative Breast Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Polly A. Niravath, MD, Principal Investigator, Medical Oncologist, The Methodist Hospital Research Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro00011685
Record Dates: First submitted 2016-06-29; First posted 2016-07-15 (Estimated); Results first posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Metastatic Triple Negative Breast Cancer
Keywords: breast cancer; nitric oxide synthase; docetaxel; L-NMMA
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — omega-N-Methylarginine; Docetaxel; Amlodipine; pegfilgrastim; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- L-NMMA 7.5 mg/kg and Docetaxel 75 mg/m2 (Experimental): Phase Ib: L-NMMA and docetaxel will be given for 6 21-day cycles. L-NMMA at doses of 7.5 mg/kg (starting dose) will be administered IV on Days 1-5. Docetaxel will be administered at 75 mg/m2 as an IV 15 min after L-NMMA infusion Day 1.
  Interventions: Drug: L-NMMA; Drug: Docetaxel; Drug: Amlodipine; Drug: Pegfilgrastim; Drug: Enteric-coated aspirin
- L-NMMA 10 mg/kg and Docetaxel 75 mg/m2 (Experimental): Phase Ib: L-NMMA and docetaxel will be given for 6 21-day cycles. L-NMMA at doses of 10 mg/kg will be administered IV on Days 1-5. Docetaxel will be administered at 75 mg/m2 as an IV 15 min after L-NMMA infusion Day 1.
  Interventions: Drug: L-NMMA; Drug: Docetaxel; Drug: Amlodipine; Drug: Pegfilgrastim; Drug: Enteric-coated aspirin
- L-NMMA 12.5 mg/kg and Docetaxel 75 mg/m2 (Experimental): Phase Ib: L-NMMA and docetaxel will be given for 6 21-day cycles. L-NMMA at doses of 12.5 mg/kg will be administered IV on Days 1-5. Docetaxel will be administered at 75 mg/m2 as an IV 15 min after L-NMMA infusion Day 1.
  Interventions: Drug: L-NMMA; Drug: Docetaxel; Drug: Amlodipine; Drug: Pegfilgrastim; Drug: Enteric-coated aspirin
- L-NMMA 15 mg/kg and Docetaxel 75 mg/m2 (Experimental): Phase Ib: L-NMMA and docetaxel will be given for 6 21-day cycles. L-NMMA at doses of 15 mg/kg will be administered IV on Days 1-5. Docetaxel will be administered at 75 mg/m2 as an IV 15 min after L-NMMA infusion Day 1.
  Interventions: Drug: L-NMMA; Drug: Docetaxel; Drug: Amlodipine; Drug: Pegfilgrastim; Drug: Enteric-coated aspirin
- L-NMMA 17.5 mg/kg and Docetaxel 100 mg/m2 (Experimental): Phase Ib: L-NMMA and docetaxel will be given for 6 21-day cycles. L-NMMA at doses of 17.5 mg/kg will be administered IV on Days 1-5. Docetaxel will be administered at 100 mg/m2 as an IV 15 min after L-NMMA infusion Day 1.
  Interventions: Drug: L-NMMA; Drug: Docetaxel; Drug: Amlodipine; Drug: Pegfilgrastim; Drug: Enteric-coated aspirin
- L-NMMA 20 mg/kg and Docetaxel 100 mg/m2 (Experimental): Phase Ib: L-NMMA and docetaxel will be given for 6 21-day cycles. L-NMMA at doses of 20 mg/kg will be administered IV on Days 1-5. Docetaxel will be administered at 100 mg/m2 as an IV 15 min after L-NMMA infusion Day 1.
  Interventions: Drug: L-NMMA; Drug: Docetaxel; Drug: Amlodipine; Drug: Pegfilgrastim; Drug: Enteric-coated aspirin
- Phase II: RP2D determined in the Phase Ib (Experimental): Phase II: L-NMMA starting dose will be the RP2D determined in the Phase Ib portion of the study.
  Interventions: Drug: L-NMMA; Drug: Docetaxel; Drug: Amlodipine; Drug: Pegfilgrastim; Drug: Enteric-coated aspirin

INTERVENTIONS:
Drug: L-NMMA — Nitric oxide synthase inhibitor
  Other Names: NG-monomethyl-l-arginine
Drug: Docetaxel — Mitotic inhibitor, cytotoxic
  Other Names: TAXOTERE
Drug: Amlodipine — Long-acting calcium channel blocker
  Other Names: besylate salt of amlodipine; NORVASC
Drug: Pegfilgrastim — Colony-stimulating factor
  Other Names: NEULASTA
Drug: Enteric-coated aspirin — non-steroidal anti-inflammatory drug
  Other Names: acetylsalicylic acid

SUMMARY:
This is a Phase Ib/II study assessing the maximum tolerated dose (MTD), dose-limiting toxicities (DLTs), recommended Phase 2 dose (RP2D), and efficacy of L-NMMA when combined with docetaxel in refractory locally advanced or metastatic triple negative breast cancer patients. The Phase Ib portion of the study is designed to investigate the combination at two dose levels of docetaxel (75 and 100 mg/m2) and 7 dose levels of L-NMMA (5, 7.5, 10, 12.5, 15, 17.5, and 20 mg/kg). The starting dose of L-NMMA will be 7.5 mg/kg. In the Phase II portion of the study, the starting dose will be the RP2D determined in the Phase Ib portion of the study.

DETAILED DESCRIPTION:
This is a Phase Ib/II study assessing the maximum tolerated dose (MTD), dose-limiting toxicities (DLTs), recommended Phase 2 dose (RP2D), and efficacy of L-NMMA when combined with docetaxel in refractory locally advanced or metastatic triple negative breast cancer patients. The Phase Ib portion of the study is designed to investigate the combination at two dose levels of docetaxel (75 and 100 mg/m2) and 7 dose levels of L-NMMA (5, 7.5, 10, 12.5, 15, 17.5, and 20 mg/kg). The starting dose of L-NMMA will be 7.5 mg/kg. L-NMMA dose will escalate/de-escalate based on DLT occurrence. For the 5, 7.5, 10, 12.5, and 15 mg/kg L-NMMA doses, docetaxel will be administered at 75 mg/m2. For the 17.5 and 20 mg/kg L-NMMA doses, docetaxel will be administered at 100 mg/m2. In the Phase II portion of the study, the starting dose will be the RP2D determined in the Phase Ib portion of the study. In the phase II portion of the study, patients will be treated with L-NMMA and taxane (docetaxel, paclitaxel, or nab-paclitaxel) per physician's choice. Patients will be treated with L-NMMA and taxane chemotherapy (docetaxel, paclitaxel, or nab-paclitaxel) per physician's choice. L-NMMA will be administered on Days 1-5 and taxane chemotherapy on Day 1 Q3W or Day 1 Q1W. L-NMMA and docetaxel will be administered at the RP2D determined in the phase Ib portion of the study. Paclitaxel at 175 mg/m2 will be IV infused over 3 hours or 80 mg/m2 will be IV infused over 1 hour, and nab-paclitaxel at 260 mg/m2 will be IV infused over 30 minutes. For L-NMMA-induced hypertension, amlodipine (10 mg) and enteric-coated low-dose aspirin (81 mg) will be orally administered. Amlodipine will be administered for 6 days at each cycle, starting 24 hours before the first dose of L-NMMA. Enteric-coated low-dose aspirin will be administered once daily during the 6 21-day cycles. For docetaxel-induced leukopenia, pegfilgrastim (6 mg) will be administered via subcutaneous injection approximately 24 hours after every dose of docetaxel.

ELIGIBILITY:
Inclusion Criteria:

Patient must meet all of the following criteria:

• Female patients with pathologically determined advanced (progressive disease or refractory to 3 cycles of standard chemotherapy) or metastatic (any line) triple negative breast cancer (TNBC). TNBC is defined as: Estrogen receptor negative and progesterone receptor negative (<10% staining by immunohistochemistry [IHC]).

Human epidermal growth factor receptor 2 (HER2) negative. HER2 negativity must be confirmed by one of the following:

* Fluorescence in situ hybridization (FISH)-negative (FISH ratio <2), or
* IHC 0-1+, or
* IHC 2+ AND FISH-negative (FISH ratio <2). Eastern Cooperative Oncology Group performance status of ≤ 2

  * Age ≥ 18 years
  * Laboratory values within the following ranges:
* Hemoglobin ≥9.0 g/dL (transfusions permitted)
* Absolute neutrophil count ≥1500/mm3 (1.5 x 109/L)
* Platelet count ≥100,000/mm3 (100 x 109/L)
* Total bilirubin <2 X upper limit of normal (ULN)
* Creatinine (Cr) <2 X ULN and Cr clearance (CrCl) ≥30 by Cockcroft and Gault
* Alanine transaminase (ALT) and aspartate transaminase (AST) <2 X ULN (if liver metastases are present then ALT and AST must be <5 X ULN)

  * Have adequate organ function (cardiac ejection fraction of ≥ 45%)
  * Negative serum pregnancy test within 7 days of the administration of the first treatment dose for women of childbearing potential (WOCBP). For WOCBP, adequate contraception must be used throughout the study.
  * Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and return for the required assessments.
  * Patient must be willing to undergo biopsies as required by the study protocol. Biopsies will be based on acceptable clinical risks as judged by investigator. Tissue from a previous biopsy will be accepted in the form of tissue slides.

Exclusion Criteria:

History of poorly controlled hypertension (defined as systolic blood pressure >150 mmHg at baseline)

* Patients with metastatic disease who have received radiation therapy, chemotherapy, or non-cytotoxic investigational agents within 2 weeks of study treatment initiation.
* Patients who received docetaxel at any line of treatment within the past 12 months
* Evidence of New York Heart Association class III or greater cardiac disease
* History of myocardial infarction, stroke, ventricular arrhythmia, or symptomatic conduction abnormality within the past 12 months
* History of congenital QT prolongation
* Absolute corrected QT interval of >480 msec in the presence of potassium >4.0 milliequivalent/L and magnesium >1.8 mg/dL
* Any medical or psychiatric condition that would prevent informed consent or limit expected survival to less than 4 weeks
* Symptomatic central nervous system metastases
* Pregnant or nursing women
* Hypersensitivity or intolerance to L-NMMA, docetaxel, amlodipine, pegfilgrastim, or their components
* Use of amlodipine or another calcium channel blocker in the past 14 days
* Alcoholism or hepatic disease with the exception of liver metastases
* Severe renal insufficiency (CrCl <30 mL/min [Cockcroft and Gault])
* History of gastrointestinal bleeding, ulceration, or perforation
* Concurrent use of potent cytochrome P450 (CYP)3A4 inhibitors
* Concurrent use of potent CYP3A4 inducers
* Concurrent use of medications that interact with nitrate/nitrites
* Use of an investigational drug within 14 days preceding the first dose of study medication.
* Concurrent use of any complementary or alternative medicines
* Patients with > Grade 2 neuropathy
* Inability to take aspirin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Polly Niravath, M.D., Principal Investigator — Houston Methodist Cancer Center
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 subjects withdrew in phase 2 and were in-evaluable.
Groups:
- Experimental: L-NMMA 7.5 mg/kg and Docetaxel 75 mg/m2: Phase Ib: L-NMMA and docetaxel will be given for 6 21-day cycles. L-NMMA at doses of 7.5 mg/kg (starting dose) will be administered IV on Days 1-5. Docetaxel will be administered at 75 mg/m2 as an IV 15 min after L-NMMA infusion Day 1.
- Experimental: L-NMMA 10 mg/kg and Docetaxel 75 mg/m2: Phase Ib: L-NMMA and docetaxel will be given for 6 21-day cycles. L-NMMA at doses of 10 mg/kg will be administered IV on Days 1-5. Docetaxel will be administered at 75 mg/m2 as an IV 15 min after L-NMMA infusion Day 1.
- Experimental: L-NMMA 12.5 mg/kg and Docetaxel 75 mg/m2: Phase Ib: L-NMMA and docetaxel will be given for 6 21-day cycles. L-NMMA at doses of 12.5 mg/kg will be administered IV on Days 1-5. Docetaxel will be administered at 75 mg/m2 as an IV 15 min after L-NMMA infusion Day 1.
- Experimental: L-NMMA 15 mg/kg and Docetaxel 75 mg/m2: Phase Ib: L-NMMA and docetaxel will be given for 6 21-day cycles. L-NMMA at doses of 15 mg/kg will be administered IV on Days 1-5. Docetaxel will be administered at 75 mg/m2 as an IV 15 min after L-NMMA infusion Day 1.
- Experimental: L-NMMA 17.5 mg/kg and Docetaxel 100 mg/m2: Phase Ib: L-NMMA and docetaxel will be given for 6 21-day cycles. L-NMMA at doses of 17.5 mg/kg will be administered IV on Days 1-5. Docetaxel will be administered at 100 mg/m2 as an IV 15 min after L-NMMA infusion Day 1.
- Experimental: L-NMMA 20 mg/kg and Docetaxel 75 mg/m2: Phase Ib: L-NMMA and docetaxel will be given for 6 21-day cycles. L-NMMA at doses of 20 mg/kg will be administered IV on Days 1-5. Docetaxel will be administered at 75 mg/m2 as an IV 15 min after L-NMMA infusion Day 1.
- Experimental: Phase II: RP2D Determined in the Phase Ib: Phase II: L-NMMA starting dose will be the RP2D determined in the Phase Ib portion of the study.
Period: Overall Study
Arm/Group | Experimental: L-NMMA 7.5 mg/kg and Docetaxel 75 mg/m2 | Experimental: L-NMMA 10 mg/kg and Docetaxel 75 mg/m2 | Experimental: L-NMMA 12.5 mg/kg and Docetaxel 75 mg/m2 | Experimental: L-NMMA 15 mg/kg and Docetaxel 75 mg/m2 | Experimental: L-NMMA 17.5 mg/kg and Docetaxel 100 mg/m2 | Experimental: L-NMMA 20 mg/kg and Docetaxel 75 mg/m2 | Experimental: Phase II: RP2D Determined in the Phase Ib
Started | 2 | 2 | 2 | 2 | 3 | 4 | 22
Evaluable Patients | 2 | 2 | 2 | 2 | 3 | 4 | 20
Completed | 0 | 0 | 0 | 1 | 0 | 1 | 4
Not Completed | 2 | 2 | 2 | 1 | 3 | 3 | 18
Not completed — Physician Decision | 2 | 1 | 2 | 1 | 1 | 2 | 12
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Complete response before the end of 6 cycles | 0 | 0 | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: 37 patients started the trial, 2 were in-evaluable from phase 2. The results are based on the 35 evaluable patients.
Groups:
- Experimental: L-NMMA 20 mg/kg and Docetaxel 100 mg/m2: Phase Ib: L-NMMA and docetaxel will be given for 6 21-day cycles. L-NMMA at doses of 20 mg/kg will be administered IV on Days 1-5. Docetaxel will be administered at 100 mg/m2 as an IV 15 min after L-NMMA infusion Day 1.
- Total: Total of all reporting groups
Arm/Group | Experimental: L-NMMA 7.5 mg/kg and Docetaxel 75 mg/m2 | Experimental: L-NMMA 10 mg/kg and Docetaxel 75 mg/m2 | Experimental: L-NMMA 12.5 mg/kg and Docetaxel 75 mg/m2 | Experimental: L-NMMA 15 mg/kg and Docetaxel 75 mg/m2 | Experimental: L-NMMA 17.5 mg/kg and Docetaxel 100 mg/m2 | Experimental: L-NMMA 20 mg/kg and Docetaxel 100 mg/m2 | Experimental: Phase II: RP2D Determined in the Phase Ib | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 3 | 4 | 20 | 35
Age, Continuous [Mean (Full Range); unit: Years] | 55 [47 to 63] | 51.5 [49 to 54] | 62 [59 to 65] | 65 [62 to 68] | 64 [56 to 80] | 63 [46 to 75] | 55 [33 to 74] | 58 [33 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 2 | 3 | 4 | 20 | 35
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Non-Hispanic Caucasian | 2 | 0 | 1 | 2 | 0 | 1 | 13 | 19
  Race: Hispanic Caucasian | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Race: African American | 0 | 2 | 0 | 0 | 2 | 2 | 6 | 12
  Race: Asian | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Stage of Breast Cancer Diagnosis [Count of Participants; unit: Participants]
  Metastatic breast cancer | 2 | 2 | 2 | 2 | 3 | 3 | 10 | 24
  Locally advanced breast cancer | 0 | 0 | 0 | 0 | 0 | 1 | 10 | 11

OUTCOME MEASURES:

1. Primary Outcome: Asses the Maximum Tolerated Dose (MTD) of L-NMMA When Combined With Docetaxel/Amlodipine in the Treatment of Refractory Locally Advanced or Metastatic TNBC Patients, Based on the Number of Dose Limiting Toxicities (DLTs) Per Dose Level.
Description: The Phase Ib portion of the study is designed to investigate the combination at two dose levels of docetaxel (75 and 100 mg/m2) and 7 dose levels of L-NMMA (5, 7.5, 10, 12.5, 15, 17.5, and 20 mg/kg). The starting dose will be L-NMMA at 7.5 mg/kg and docetaxel at 75 mg/m2. As patients are accrued, a standard Bayesian model averaging continual reassessment method (CRM) approach will be used to determine the appropriate dosage. For a dose level to be chosen as the MTD, at least 4 patients must have received said dose without experiencing a significant number of DLTs based on the Bayesian Model Averaging Continual Reassessment Method.
Time Frame: DLTs assessment window is the duration required for completing one full cycle (through Day 21).
Population: 15 participants participated in Phase Ib portion of the trial until the MTD was determined after 4 patient completed at least one cycle of treatment at the same dose without DLTs.
Measure: Number; unit: mg/kg
Groups:
- Phase Ib - Dose Finding - L-NMMA: The Phase Ib portion of the study is designed to investigate the combination at two dose levels of docetaxel (75 and 100 mg/m2) and 7 dose levels of L-NMMA (5, 7.5, 10, 12.5, 15, 17.5, and 20 mg/kg). The starting dose will be L-NMMA at 7.5 mg/kg and docetaxel at 75 mg/m2.
Arm/Group | Phase Ib - Dose Finding - L-NMMA
Number analyzed (Participants) | 15
mg/kg | 20

2. Primary Outcome: Clinical Benefit Rate
Description: Primary Outcome Measure for Phase II: Determine the number of participants with complete response, partial response, or stable disease after 6 cycles of L-NMMA combined with taxane chemotherapy (docetaxel, paclitaxel, or nab-paclitaxel)/amlodipine, as assessed by the RECIST 1.1.
  * CR (complete response) = disappearance of all target lesions
  * PR (partial response) = 30% decrease in the sum of the longest diameter of target lesions
  * PD (progressive disease) = 20% increase in the sum of the longest diameter of target lesions
  * SD (stable disease) = small changes that do not meet above criteria
  * Treatment Failure: taken off the study because of adverse events before the first restaging scan after cycle 2
Time Frame: The approximate length of the study from Cycle 1, Day 1 will be approximately seven months (approximately four months of treatment plus three months of follow-up).
Population: 24 subjects participated in the Phase II portion of the trial
Measure: Count of Participants; unit: Participants
Groups:
- Experimental: Phase Ib: L-NMMA and docetaxel will be given for 6 21-day cycles. L-NMMA at doses of 5, 7.5 (starting dose), 10, 12.5, 15, 17.5, and 20 mg/kg will be administered IV on Days 1-5. For 5-15 mg/kg L-NMMA doses, docetaxel will be administered at 75 mg/m2. For 17.5 and 20 mg/kg L-NMMA doses, docetaxel will be administered at 100 mg/m2. Docetaxel will be administered IV 15 min after the Day 1 L-NMMA infusion. Amlodipine (10 mg) will be orally administered daily for 6 days, starting 24 hours before the Day 1 L-NMMA infusion. Enteric-coated aspirin (81 mg) will be orally administered once daily during the 6 21-day cycles. Pegfilgrastim (6 mg) will be administered subcutaneously 24 h after docetaxel.
  Phase II: L-NMMA starting dose will be the RP2D determined in the Phase Ib portion of the study.
  L-NMMA: Nitric oxide synthase inhibitor
  Docetaxel: Mitotic inhibitor, cytotoxic
  Amlodipine: Long-acting calcium channel blocker
  Pegfilgrastim: Colony-stimulating factor
  Enteric-coated aspirin: non-steroidal anti-inflammatory drug
Arm/Group | Experimental
Number analyzed (Participants) | 24
Participants
  Metastatic breast cancer: number analyzed (Participants) | 13
  Metastatic breast cancer: Complete Response | 0
  Metastatic breast cancer: Partial Response | 2
  Metastatic breast cancer: Stable Disease | 3
  Metastatic breast cancer: Progressive Disease | 6
  Metastatic breast cancer: Treatment Failure | 2
  Locally advanced breast cancer: number analyzed (Participants) | 11
  Locally advanced breast cancer: Complete Response | 4
  Locally advanced breast cancer: Partial Response | 5
  Locally advanced breast cancer: Stable Disease | 1
  Locally advanced breast cancer: Progressive Disease | 1
  Locally advanced breast cancer: Treatment Failure | 0

3. Secondary Outcome: Dose Limiting Toxicities (DLTs) and Other Adverse Events
Description: Describe the DLTs and other adverse events associated with L-NMMA when combined with docetaxel/amlodipine, as assessed by the CTCAE v4.03 Any Grade ≥ 3 Adverse Events (AE) unless there is clear alternative evidence that the AE was not caused by the study treatment.
Time Frame: as for outcome 2
Population: Patients who experienced adverse events Grade ≥ 3
Measure: Count of Units; unit: Grade ≥ 3 AE
Units Other Than Participants: Grade ≥ 3 AE
Arm/Group | Experimental: L-NMMA 7.5 mg/kg and Docetaxel 75 mg/m2 | Experimental: L-NMMA 10 mg/kg and Docetaxel 75 mg/m2 | Experimental: L-NMMA 12.5 mg/kg and Docetaxel 75 mg/m2 | Experimental: L-NMMA 15 mg/kg and Docetaxel 75 mg/m2 | Experimental: L-NMMA 17.5 mg/kg and Docetaxel 100 mg/m2 | Experimental: L-NMMA 20 mg/kg and Docetaxel 100 mg/m2 | Experimental: Phase II: RP2D Determined in the Phase Ib
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 3 | 4 | 20
Number analyzed (Grade ≥ 3 AE) | 0 | 1 | 0 | 0 | 7 | 3 | 3
Grade ≥ 3 AE
  Constitutional | 0 | 0 | 0 | 0 | 2 | 1 | 0
  Peripheral neuropathy | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Dermatological | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Infectious | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Renal | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Elevation of AST/ALT | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dehydration | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Gastric | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Cardiac | 0 | 0 | 0 | 0 | 2 | 0 | 1
  Vascular | 0 | 0 | 0 | 0 | 1 | 0 | 0

4. Secondary Outcome: Recommended Phase 2 Dose (RP2D) of the L-NMMA and Docetaxel Combination
Description: Determine the RP2D of the L-NMMA and docetaxel combination based on the occurrence of DLTs during Phase Ib portion of the study.
  As patients are accrued, they will start with 7.5 mg/kg of L-NMMA and 75 mg/m2 of docetaxel and their DLTs will be assessed after completion of the first cycle. This will determine the next cohort dose, until at least 4 patients receive the dose with minimal DLTs that won't require dose reduction.
Time Frame: The Dose Limiting Toxicities (DLT) assessment window is the duration required for completing one full cycle (through Day 21).
Population: as for outcome 1
Measure: Number; unit: mg/kg
Arm/Group | Phase Ib - Dose Finding - L-NMMA
Number analyzed (Participants) | 15
mg/kg | 20

5. Secondary Outcome: Antitumor Activity
Description: Assess the antitumor activity of L-NMMA when combined with taxane chemotherapy (docetaxel, paclitaxel, or nab-paclitaxel)/amlodipine, as assessed by the RECIST 1.1.
  * CR (complete response) = disappearance of all target lesions
  * PR (partial response) = 30% decrease in the sum of the longest diameter of target lesions
  * PD (progressive disease) = 20% increase in the sum of the longest diameter of target lesions
  * SD (stable disease) = small changes that do not meet above criteria
  * Treatment Failure: taken off the study because of adverse events before the first restaging scan after cycle 2
Time Frame: as for outcome 2
Population: 22 subjects participated in the Phase II portion of the trial (2 patients were in-evaluable) 4 subjects were included from Phase Ib portion who received the same dose.
Measure: Count of Participants; unit: Participants
Groups:
- Experimental: Phase II: RP2D Determined in the Phase Ib: Phase II: L-NMMA starting dose will be the RP2D determined in the Phase Ib portion of the study.
  L-NMMA and docetaxel will be given for 6 21-day cycles. L-NMMA at doses of 20 mg/kg will be administered IV on Days 1-5. Docetaxel will be administered at 100 mg/m2 as an IV 15 min after L-NMMA infusion Day 1.
Arm/Group | Experimental: L-NMMA 7.5 mg/kg and Docetaxel 75 mg/m2 | Experimental: L-NMMA 10 mg/kg and Docetaxel 75 mg/m2 | Experimental: L-NMMA 12.5 mg/kg and Docetaxel 75 mg/m2 | Experimental: L-NMMA 15 mg/kg and Docetaxel 75 mg/m2 | Experimental: L-NMMA 17.5 mg/kg and Docetaxel 100 mg/m2 | Experimental: L-NMMA 20 mg/kg and Docetaxel 100 mg/m2 | Experimental: Phase II: RP2D Determined in the Phase Ib
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 3 | 4 | 20
Participants
  Complete Response (100% reduction) | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Partial Response (<100% reduction) | 0 | 0 | 0 | 1 | 0 | 1 | 7
  Stable Disease (< 20% change) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Progressive Disease (> 20% growth) | 2 | 1 | 2 | 1 | 1 | 2 | 7
  Treatment Failure | 0 | 1 | 0 | 0 | 2 | 1 | 2

6. Secondary Outcome: Time to Maximum Plasma Concentration of L-NMMA and Docetaxel
Description: Determine the time to maximum plasma concentration of the L-NMMA and docetaxel combination.
Time Frame: Blood samples will be collected predose (10-30 minutes before L-NMMA infusion) on Days 1, 2, and 5 of Cycle 1 and Days 1 and 5 of Cycle 2 for determination of L-NMMA plus docetaxel plasma PK.
Population: To determine the PK of L-NMMA, we assayed serum samples from two patients receiving L-NMMA at 15 mg/kg and docetaxel at 75 mg/m2 and two patients receiving L-NMMA at 17.5 mg/kg and docetaxel at 100 mg/m2.
Measure: Mean (Full Range); unit: Hours
Arm/Group | Experimental: L-NMMA 15 mg/kg and Docetaxel 75 mg/m2 | Experimental: L-NMMA 17.5 mg/kg and Docetaxel 100 mg/m2
Number analyzed (Participants) | 2 | 2
Hours
  Tmax for LNMMA | 2 [0 to 24] | 2 [0 to 24]
  Tmas for Docetaxel | 4 [0 to 30] | 4 [0 to 30]

7. Other Pre Specified Outcome: Area Under the Plasma Concentration Curve of the L-NMMA and Docetaxel Combination
Description: Determine the area under the plasma concentration curve of the L-NMMA and docetaxel combination
Time Frame: 18 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Predictive Biomarkers
Description: Determine potential predictive biomarkers including serum levels of nitrate/nitrite; serum levels of inflammatory biomarkers; angiogenesis-related biomarkers; and RPL39, MLF2, and phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha (PIK3CA) mutations in cell-free DNA
Time Frame: 18 weeks
Reporting Status: Not Posted

9. Primary Outcome: Asses the Maximum Tolerated Dose (MTD) of Docetaxel When Combined With L-NMMA/Amlodipine in the Treatment of Refractory Locally Advanced or Metastatic TNBC Patients, Based on the Number of Dose Limiting Toxicities (DLTs) Per Dose Level.
Description: as for outcome 1
Time Frame: DLTs assessment window is the duration required for completing one full cycle (through Day 21).
Population: as for outcome 1
Measure: Number; unit: mg/m^2
Groups:
- Phase Ib - Dose Finding - Docetaxel: The Phase Ib portion of the study is designed to investigate the combination at two dose levels of docetaxel (75 and 100 mg/m2) and 7 dose levels of L-NMMA (5, 7.5, 10, 12.5, 15, 17.5, and 20 mg/kg). The starting dose will be L-NMMA at 7.5 mg/kg and docetaxel at 75 mg/m2.
Arm/Group | Phase Ib - Dose Finding - Docetaxel
Number analyzed (Participants) | 15
mg/m^2 | 100

10. Secondary Outcome: Recommended Phase 2 Dose (RP2D) of the L-NMMA and Docetaxel Combination
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Number; unit: mg/m^2
Arm/Group | Phase Ib - Dose Finding - Docetaxel
Number analyzed (Participants) | 15
mg/m^2 | 100

ADVERSE EVENTS:
Time Frame: From informed consent signing up to and including 30 days after the last treatment dose. All patients will be followed for 3 months after the final dose of treatment and will be evaluated accordingly with the required standard of care labs and tests. All reported events are included when the subjects was on study, or within the follow up period, up to 3 months after the final dose. A maximum duration of 8 months.
Groups:
- Experimental: L-NMMA 7.5 mg/kg and Docetaxel 75 mg/m2: Phase Ib: L-NMMA and docetaxel will be given for 6 21-day cycles. L-NMMA at doses of 7.5 mg/kg (starting dose) will be administered IV on Days 1-5. Docetaxel will be administered at 75 mg/m2 as an IV 15 min after L-NMMA infusion Day 1.
  Amlodipine: Long-acting calcium channel blocker
  Pegfilgrastim: Colony-stimulating factor
  Enteric-coated aspirin: non-steroidal anti-inflammatory drug
Arm/Group | Experimental: L-NMMA 7.5 mg/kg and Docetaxel 75 mg/m2 | Experimental: L-NMMA 10 mg/kg and Docetaxel 75 mg/m2 | Experimental: L-NMMA 12.5 mg/kg and Docetaxel 75 mg/m2 | Experimental: L-NMMA 15 mg/kg and Docetaxel 75 mg/m2 | Experimental: L-NMMA 17.5 mg/kg and Docetaxel 100 mg/m2 | Experimental: L-NMMA 20 mg/kg and Docetaxel 100 mg/m2 | Experimental: Phase II: RP2D Determined in the Phase Ib
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2 | 0/3 | 0/4 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/2 | 2/2 | 0/2 | 0/2 | 1/3 | 1/4 | 3/20
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 2/2 | 1/2 | 3/3 | 4/4 | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: L-NMMA 7.5 mg/kg and Docetaxel 75 mg/m2 (N=2) | Experimental: L-NMMA 10 mg/kg and Docetaxel 75 mg/m2 (N=2) | Experimental: L-NMMA 12.5 mg/kg and Docetaxel 75 mg/m2 (N=2) | Experimental: L-NMMA 15 mg/kg and Docetaxel 75 mg/m2 (N=2) | Experimental: L-NMMA 17.5 mg/kg and Docetaxel 100 mg/m2 (N=3) | Experimental: L-NMMA 20 mg/kg and Docetaxel 100 mg/m2 (N=4) | Experimental: Phase II: RP2D Determined in the Phase Ib (N=20)
Change in mental status (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Change in mental status (due to multiple brain mets & possible leptomeningeal disease)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Right upper extremity Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — A disorder characterized by an infectious process involving the skin such as cellulitis.
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute renal insufficiency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest wall significant Erythema on front and back (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — L. Chest wall-Significant Erythema on front and back, Skin peeling and hardness of chest wall
Clinical sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: L-NMMA 7.5 mg/kg and Docetaxel 75 mg/m2 (N=2) | Experimental: L-NMMA 10 mg/kg and Docetaxel 75 mg/m2 (N=2) | Experimental: L-NMMA 12.5 mg/kg and Docetaxel 75 mg/m2 (N=2) | Experimental: L-NMMA 15 mg/kg and Docetaxel 75 mg/m2 (N=2) | Experimental: L-NMMA 17.5 mg/kg and Docetaxel 100 mg/m2 (N=3) | Experimental: L-NMMA 20 mg/kg and Docetaxel 100 mg/m2 (N=4) | Experimental: Phase II: RP2D Determined in the Phase Ib (N=20)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Acute allergic reaction (Immune system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bicytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bilateral Leg Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Body Aches (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 7 (7)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Contusion (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Decreased Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 6 (7)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated AST and ALT (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fatigue and weakness (General disorders) | 1 (3) | 1 (1) | 1 (1) | 1 (1) | 2 (4) | 1 (1) | 5 (6)
Gum bleeding (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand-foot Syndrome (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 8 (8)
Arm and shoulder swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower abdomen incision packing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Narrowing of brachiocephalic vein stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Oral mucositis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sensitivity to light (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomitting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Weight loss (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/03/NCT02834403/Prot_SAP_000.pdf